CLINICAL TRIAL: NCT01617707
Title: Safe and Effective Sedation in Chronic Alcoholic Patients Underwent Diagnostic Endoscopic Procedures: a Prospective, Randomized Study Comparing Midazolam and Propofol With Midazolam
Brief Title: Safe and Effective Sedation in Chronic Alcoholic Patients Underwent Diagnostic Endoscopic Procedures: Study Comparing Midazolam and Propofol With Midazolam
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because of difficulties for participants enrollment
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2012-0181
Record Dates: First submitted 2012-06-01; First posted 2012-06-12 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2014-03

CONDITIONS: Chronic Alcoholism
Keywords: sedation; endoscopy; midazolam; propofol; chronic alcoholics
MeSH Terms: conditions — Alcoholism | interventions — Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional sedation group (Active Comparator): midazolam
  Interventions: Drug: Midazolam
- BPS group (Experimental): midazolam plus propofol
  Interventions: Drug: Midazolam plus propofol

INTERVENTIONS:
Drug: Midazolam plus propofol — In both study arms, patients who were 20-70 years of age received an initial intravenous bolus of 0.05mg/kg of midazolam, while patients ≥71 years of age received an initial intravenous dose of 1mg of midazolam. After 2min following this initial dose of midazolam, the conventional sedation group received additional boluses as needed of 1 to 2 mg of midazolam at the discretion of the endoscopist, to target moderate sedation. The BPS group received an initial 0.5mg/kg bolus of intravenous propofol at 2min after midazolam administration. Subsequent incremental boluses of 10 to 20 mg of propofol were allowed to be given at the discretion of the endoscopist every 30s to target moderate sedation.
  Arms: BPS group
Drug: Midazolam — In both study arms, patients who were 20-70 years of age received an initial intravenous bolus of 0.05mg/kg of midazolam, while patients ≥71 years of age received an initial intravenous dose of 1mg of midazolam. After 2min following this initial dose of midazolam, the conventional sedation group received additional boluses as needed of 1 to 2 mg of midazolam at the discretion of the endoscopist, to target moderate sedation. The BPS group received an initial 0.5mg/kg bolus of intravenous propofol at 2min after midazolam administration. Subsequent incremental boluses of 10 to 20 mg of propofol were allowed to be given at the discretion of the endoscopist every 30s to target moderate sedation.
  Arms: conventional sedation group

SUMMARY:
Sedative endoscopic examination using sedative premedication has been undertaken to induce conscious sedation for comfortable and painless endoscopy. Midazolam has been most widely used as a sedative premedication because it has lots of advantages, such as a short half-life, a faster onset of sedation and an excellent sedative hypnotic effect. However, midazolam has been used regardless of whether or not alcohol although using midazolam in chronic alcoholics is related to paradoxical reaction, characterized by increased talkativeness, emotional release, excitement, and excessive movement. In recent years, propofol has been used safety and effectively in sedative GI endoscopy because of its potent hypnotic effect and its ultrashort pharmacokinetic profile. Therefore, The present study was conducted to compare the safety and efficacy of BPS (propofol in combination with midazolam) with conventional sedation (midazolam) in chronic alcoholic patients undergoing diagnostic GI endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20
* ECOG ≥ 2
* patient who consents to enroll the trial

Exclusion Criteria:

* age < 20
* pregnant or lactating women
* American Society of Anesthesiology (ASA) physical status class V
* chronic pulmonary disease
* history of allergic to propofol
* history of complication of sedation endoscope
* liver failure or hepatic encephalopathy
* who didn't consented to enroll the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction of endoscopists, nurses and patients | about 5 minutes after the end of the procedure
  endoscopists and nurses - about 5 minutes after the end of the procedure / patients - upon meeting discharge criteria (modified Aldrete score), an expected average of 20min

SECONDARY OUTCOMES:
completion rate of endoscopy | about 5 minutes after the end of procedure
number of participants with complications | participants will be followed during the procedure and recovery time, an expected average of 20 min
  hypoxemia (SpO2<90%), hypotension (SBP<90mmHg), bradycardia (HR<50/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea